CLINICAL TRIAL: NCT01878422
Title: SEQUENTIAL TREATMENT STRATEGY FOR METASTATIC COLORECTAL CANCER: A PHASE III PROSPECTIVE RANDOMIZED MULTICENTER STUDY OF CHEMOTHERAPY (CT) WITH OR WITHOUT BEVACIZUMAB AS FIRST-LINE THERAPY FOLLOWED BY TWO PHASE III RANDOMIZED STUDIES OF CT ALONE OR CT PLUS BEVACIZUMAB WITH OR WITHOUT CETUXIMAB AS SECOND-LINE THERAPY
Brief Title: Sequential Treatment Strategy for Metastatic Colorectal Cancer
Acronym: ITACa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST153.01; 2007-004539-44 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-17 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm A: FOLFIRI or FOLFOX + Bevacizumab (Experimental): * BEVACIZUMAB: Day 1,1st cycle 5 mg/kg IV infusion of 90 min Day 1, 2nd cycle if well tolerated, 5 mg/kg IV infusion of 60 min Day 1, 3rd cycle and subsequent cycles if well tolerated, 5 mg/kg IV infusion of 30 min after 5-FU bolus
  * FOLFIRI Day 1: Irinotecan 180 mg/m2 IV infusion 30-90 min
  Day 1,2:
  L-Folinic acid 100 mg/m2 IV infusion of 2 hours 5-Fluorouracil 400 mg/m2 as a bolus 5-Fluorouracil 600 mg/m2 continuous IV infusion of 22 hours
  - FOLFOX Day 1: Oxaliplatin 85 mg/m2 IV infusion of 2hours
  Day 1,2:
  L-Folinic acid 100 mg/m2 IV infusion of 2 hours 5-Fluorouracil 400 mg/m2 as a bolus 5-Fluorouracil 600 mg/m2 continuous IV infusion of 22 hours
  Interventions: Drug: Arm A: FOLFIRI or FOLFOX + Bevacizumab
- Arm B: FOLFIRI or FOLFOX (Experimental): If FOLFIRI: FOLFIRI as specified in arm A without Bevacizumab If FOLFOX: FOLFOX as specified in arm A without Bevacizumab
  Interventions: Drug: Arm B: FOLFIRI or FOLFOX
- Arm C: FOLFIRI or FOLFOX (Experimental): Arm C: FOLFIRI or FOLFOX: for patients from arm A: FOLFIRI or FOLFOX (the CT schedule not received in 1st line trial, as defined in arm B)
  Interventions: Drug: Arm B: FOLFIRI or FOLFOX
- Arm D: FOLFIRI or FOLFOX plus CETUXIMAB (Experimental): Arm D: FOLFIRI or FOLFOX plus CETUXIMAB: for patients from arm B: FOLFIRI or FOLFOX (the CT schedule not received in 1st line trial, as described in arm B) plus CETUXIMAB
  Interventions: Drug: Arm D: FOLFIRI or FOLFOX plus CETUXIMAB
- Arm E: FOLFIRI or FOLFOX plus BEVACIZUMAB (Experimental): for patients from arm B: FOLFIRI or FOLFOX (the CT schedule not received in the 1st line trial, as defined in arm B) plus BEVACIZUMAB
  Interventions: Drug: Arm A: FOLFIRI or FOLFOX + Bevacizumab
- Arm F: FOLFIRI or FOLFOX plus BEVACIZUMAB and CETUXIMAB; (Experimental): for patients from arm B: FOLFIRI or FOLFOX (the CT schedule not received in the first-line trial, as defined in arm B) plus BEVACIZUMAB and CETUXIMAB; cycle to be repeated every 2 weeks, whilst cetuximab will be administered weekly.
  Interventions: Drug: Arm F: FOLFIRI or FOLFOX plus BEVACIZUMAB and CETUXIMAB

INTERVENTIONS:
Drug: Arm A: FOLFIRI or FOLFOX + Bevacizumab — Arm A: FOLFIRI or FOLFOX + Bevacizumab or Arm E: FOLFIRI or FOLFOX plus BEVACIZUMAB
  Other Names: Arm E: FOLFIRI or FOLFOX plus BEVACIZUMAB
  Arms: Arm A: FOLFIRI or FOLFOX + Bevacizumab; Arm E: FOLFIRI or FOLFOX plus BEVACIZUMAB
Drug: Arm B: FOLFIRI or FOLFOX — Arm B: FOLFIRI or FOLFOX or Arm C: FOLFIRI or FOLFOX
  Other Names: Arm C: FOLFIRI or FOLFOX
  Arms: Arm B: FOLFIRI or FOLFOX; Arm C: FOLFIRI or FOLFOX
Drug: Arm D: FOLFIRI or FOLFOX plus CETUXIMAB — Arm D: FOLFIRI or FOLFOX plus CETUXIMAB
  Other Names: FOLFIRI or FOLFOX plus CETUXIMAB
  Arms: Arm D: FOLFIRI or FOLFOX plus CETUXIMAB
Drug: Arm F: FOLFIRI or FOLFOX plus BEVACIZUMAB and CETUXIMAB — Arm F: FOLFIRI or FOLFOX plus BEVACIZUMAB and CETUXIMAB
  Other Names: FOLFIRI or FOLFOX plus BEVACIZUMAB and CETUXIMAB
  Arms: Arm F: FOLFIRI or FOLFOX plus BEVACIZUMAB and CETUXIMAB;

SUMMARY:
Study Design: This is a pragmatic study on the management strategy for patients with metastatic colorectal cancer (CRC) who are candidates for CT, independently of any previous adjuvant therapy received. The aim of this study is to define the role of new target molecules in combination with CT in first- and second line treatment.

First line study: Eligible patients were randomized to either treatment:

Arm A: FOLFIRI or FOLFOX + Bevacizumab, cycle to be repeated every 2 weeks

* BEVACIZUMAB: Day 1,1st cycle 5 mg/kg IV infusion of 90 min Day 1, 2nd cycle if well tolerated, 5 mg/kg IV infusion of 60 min Day 1, 3rd cycle and subsequent cycles if well tolerated, 5 mg/kg IV infusion of 30 min after 5-Fluorouracile (FU) bolus
* FOLFIRI Day 1: Irinotecan 180 mg/m2 IV infusion 30-90 min

Day 1,2:

L-Folinic acid 100 mg/m2 IV infusion of 2 hours 5-Fluorouracil 400 mg/m2 as a bolus 5-Fluorouracil 600 mg/m2 continuous IV infusion of 22 hours - FOLFOX Day 1: Oxaliplatin 85 mg/m2 IV infusion of 2hours

Day 1,2:

L-Folinic acid 100 mg/m2 IV infusion of 2 hours 5-Fluorouracil 400 mg/m2 as a bolus 5-Fluorouracil 600 mg/m2 continuous IV infusion of 22 hours Arm B: FOLFIRI or FOLFOX, cycle to be repeated every 2 weeks If FOLFIRI: FOLFIRI as specified in arm A without Bevacizumab If FOLFOX: FOLFOX as specified in arm A without Bevacizumab Duration of Therapy For both arms, CT was repeated until progressive disease (PD) or unacceptable toxicity occurs. If unacceptable CT-related toxicity occurs in ARM A, in the absence of PD patients stopped CT and continued with only bevacizumab 5 mg/kg as a 30-min infusion every 2 weeks until progression or intolerable toxicity occurred.

Second line - it is divided in two different studies (2A and 2B):

Study 2A: Patients from arm A and Kras Wild Type were randomized to:

* Arm C: FOLFIRI or FOLFOX (the CT schedule not received in 1st line trial, as defined in arm B)
* Arm D: FOLFIRI or FOLFOX (the CT schedule not received in 1st line trial, as described in arm B) plus CETUXIMAB CETUXIMAB 1st cycle Day 1 400 mg/m2 infusion of 120 min 2 hrs before CT infusion 1st cycle Day 8 and subsequent cycles 250 mg/m2 infusion of 60 min 1 hr before CT infusion Patients from arm A and Kras Mutant were treated according to arm C.

Study 2B: Patients from arm B and Kras Wild Type were randomized to:

* Arm E: FOLFIRI or FOLFOX (the CT schedule not received in the 1st line trial, as defined in arm B) plus BEVACIZUMAB
* Arm F: FOLFIRI or FOLFOX (the CT schedule not received in the first-line trial, as defined in arm B) plus BEVACIZUMAB and CETUXIMAB; cycle to be repeated every 2 weeks, whilst cetuximab will be administered weekly.
* BEVACIZUMAB 2nd day of 1st cycle 5 mg/kg IV infusion of 90 min 2nd day of 2 nd cycle if well tolerated, 5 mg/kg IV infusion of 60 min 2nd day of 3 rd cycle and subsequent cycles if well tolerated, 5 mg/kg IV infusion of 30 min after the end of 5-FU bolus on the 2nd day
* CETUXIMAB 1st cycle Day 1 400 mg/m2 infusion of 120 min 2 hr before CT infusion 1st cycle Day 8 and subsequent cycles 250 mg/m2 infusion of 60 min 1 hr before CT infusion If cetuximab will be stopped for any of the reasons specified in this protocol, bevacizumab will be administered as defined in arm A of the 1st line study Patients from arm B and Kras Mutant were treated according to arm E. Objectives of study The primary objective of the 1st line study is to determine whether the addition of bevacizumab to a poly-chemotherapy (polyCT) regimen (FOLFIRI or FOLFOX) improves efficacy in terms of progression-free survival (PFS). The secondary objectives of the 1st line study are to determine the Overall Response Rate (ORR) and the safety profile of the treatments administered.

The primary objective of the 2nd line studies is to determine, separately for each study, whether the addition of cetuximab to a polyCT schemes (FOLFOX or FOLFIRI), or to polyCT schemes plus bevacizumab, improves efficacy in terms of PFS.The secondary objectives of the 2nd line studies are to determine the ORR, the overall survival (OS) and the safety profile of the treatments administered.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed untreated metastatic or locally advanced, non resectable CRC; previous adjuvant chemotherapy for CRC or neoadjuvant/adjuvant chemoradiotherapy for rectal cancer is permitted but must have been completed at least 6 months prior to enrolment;
2. Resected CRC patients who have developed metastases do not require separate histological or cytological confirmation unless > 5 yrs have elapsed between primary surgery or primary tumor stage I;
3. Evaluation of Kras status from the primary tumor or metastases
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST criteria)
5. Age ≥ 18 years and < 70 years with Performance Status (ECOG) ≤ 2 or age > 70 years with ECOG ≤ 1;
6. Estimated life expectancy of at least 12 weeks;
7. Adequate hematological, hepatic and renal function, as follows: hemoglobin ≥ 9 g/dl,absolute neutrophil count ≥1,500/μL, platelets ≥100,000/μL, total bilirubin ≤1.5 x upper limit of normal (ULN),alkaline phosphatase, aspartate aminotransferase (AST(SGOT)) and alanine aminotransferase (ALT(SGPT)) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases present), serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance >50 mL/min (calculated on the basis of Standard Cockcroft and Gault Formula, urinary excretion (if protein > 30 mg/dL or +1, patients must have ≤ 1 g of protein/24 hours)
8. Either international normalized ratio (INR) or activated partial thromboplastin time (APTT) < 1.5 x ULN and D-dimer within normal range (if abnormal, thromboembolic events must be excluded);
9. Negative pregnancy test no more than 7 days before randomization; test pregnancy can be omitted only in women without any reproductive potential (e.g.: postmenopausal women, i.e. amenorrhoea ≥2 years or with previous hysterectomy or bilateral ovariectomy). Women of child-bearing potential and men must agree to use adequate contraception at the time of randomization and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician and coordinating centre (CC) immediately; women in lactation period must be excluded;
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior treatment with cetuximab, bevacizumab or other anti Epidermal Growth Factor Receptor (antiEGFR) or anti-angiogenesis agents;
2. Prior chemotherapy or immunotherapy for metastatic or advanced disease;
3. Participation in another clinical trial with any investigational agents ≤ 30 days prior to study randomization;
4. Contraindications or hypersensitivity to study drugs;
5. Treatment with other concomitant antineoplastic drugs;
6. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma and in situ carcinoma of the uterine cervix);
7. Symptomatic brain or central nervous system metastases or clinically relevant central nervous diseases (for example: primary brain tumor, uncontrolled convulsions with medical therapy, carcinomatous meningitis);
8. Grade > 1 peripheral neuropathy (as defined by the National Cancer Institute - Common Toxicity Criteria for Adverse Effects (NCI CTCAE) v3.0);
9. Clinically significant (i.e. active) cardiovascular disease e.g. cerebrovascular accidents ≤ 6 months prior to randomization), myocardial infarction (≤ 1 year prior to randomization), uncontrolled hypertension whilst receiving chronic medication, unstable angina, New York Heart Association (NYHA) grade II or more congestive heart failure,or serious cardiac arrhythmia requiring medication;
10. Malabsorption syndrome or lack of physical integrity of the gastrointestinal tract. Diverticulitis. Patients with colostomy or ileostomy may enter at the investigator's discretion. History of trachea-oesophageal fistula or any other type of fistula (e.g. abdominal), gastrointestinal perforation, intra-abdominal abscess;
11. Interstitial pneumonia or extensive symptomatic fibrosis of the lungs;
12. Serious, non-healing wound, ulcer, or bone fracture; significant traumatic injury in the 4 weeks prior to enrolment (complete recover must have occurred);
13. Major surgery (e.g. laparotomy) in the 4 weeks prior to study randomization;
14. Minor surgery in the 2 weeks prior to study randomization. Insertion of a central vascular access device for chemotherapy infusion must be done at least 2 days prior to the start of treatment. Patients will be randomized only if they have recovered from all surgery related toxicities;
15. Bleeding diathesis or coagulopathy;
16. Pulmonary embolism or any arterial thromboembolism;
17. Deep vein thrombosis or other significant thromboembolic event;
18. Clinically significant peripheral vascular disease;
19. Previous organ transplantation that requires immunosuppressive therapy;
20. Need for chronic oral steroid use ( ≥10 mg/day of methylprednisolone or equivalent) for the treatment of a nonmalignant condition other than intermittent prophylactic use as an antiemetic and inhaled steroid use;
21. Chronic use of aspirin (> 325 mg/day) or other non steroidal anti-inflammatory agents (those known to inhibit platelet function at doses used to treat chronic inflammatory diseases);
22. In treatment with antiplatelets agents (i.e clopidogrel > 75 mg/day, ticlopidine,dipyridamole);
23. Undergoing treatment with sorivudine or its chemically-related analogues (such as brivudine);
24. Full-dose oral or parenteral anticoagulants or thrombolytic treatment for therapeutic purposes ≤10 days prior to study randomization;
25. Geographic inaccessibility;
26. Any radiation therapy completed ≤ 4 weeks prior to study randomization. If the radiated lesion/s is/are the only site of disease, and if it/they show progression after the radiotherapeutic procedure, the patient will become eligible for the study;
27. Previous embolization or thermoablation of metastases ≤ 30 days prior to study randomization. If these lesions are the only site of disease, and if they show progression after the embolization or thermoablation procedure, the patient will become eligible for the study;
28. Laboratory abnormality or medical or psychiatric disorders that would interfere with informed consent or compliance, or which could indicate a contraindication to patient enrolment into the study (also known dihydropyrimidine dehydrogenase deficit);
29. HIV-positivity, whether or not symptomatic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2007-11; Primary Completion 2014-03 (Actual); Study Completion 2016-06-11 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) of first and second line treatment strategy | 6 years
  To compare the Progression Free Survival (PFS) between different treatment arms in patients of first line treatment and, subsequently, the same analisys will be performed in patients treated in second line therapy.

SECONDARY OUTCOMES:
Overal Response Rate (ORR) of first and second line treatment strategy | 6 years
  To compare the Overal Response Rate (ORR) between different treatment arms in patients of first line treatment and, subsequently, the same analisys will be performed in patients treated in second line therapy.
Overal Survival (OS) of second line treatment | 6 years
  To compare the Overal Survival (OS) between different treatment arms in patients of second line treatment
Number of partecipants with adverse events as a measure of safety and tolerability | 6 years
  To compare the number of partecipants with adverse events as a measure of safety and tolerability between different treatment arms of first line treatment and, subsequently, the same analisys will be performed in patients treated in second line therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dino Amadori, Principal Investigator — IRST IRCCS, Meldola
Locations (23):
- Italy (23):
  - Dipartimento Oncologia Ematologia - Policlinico S.Orsola-Malpighi - Università di Bologna, Bologna, BO
  - Ist. di Ematologia e Oncologia Medica "L. e A. Seragnoli" - Università di Bologna, Bologna, BO
  - Ospedale Bellaria-Maggiore, AUSL Città di Bologna, Bologna, BO
  - P.O. San lazzaro, Alba, CN
  - Ospedale Buffalini - ASL Cesena, Cesena, FC
  - Irccs Irst, Meldola (FC), FC
  - Azienda Ospedaliero - Università di Ferrara, Ferrara, FE
  - Ospedale Vito Fazzi, Lecce, LE
  - Ospedale Ramazzini - ASL Modena, Carpi, MO
  - Centro Oncologico Modenese - Policlinico di Modena, Modena, MO
  - Ospedale degli Infermi - AUSL di Ravenna, Faenza, RA
  - Ospedale Civile di Lugo -AUSL di Ravenna, Lugo, RA
  - Ospedale S.Maria delle Croci, Ravenna, RA
  - ospedale Civile Cattolica, Cattolica, RN
  - Ospedale Infermi - Azienda USL di Rimini, Rimini, RN
  - AOU S.Giovanni Battista di Torino (Molinette) Presidio San Lazzaro, Torino, TO
  - Azienda Sanitaria Ospedaliera S. Giovanni Battista - Molinette, Torino, TO
  - Ospedale Cardinal Massaia, Asti
  - Azienda ULSS 1 di Belluno, Belluno
  - Ospedale A.Perrino, Brindisi
  - Azienda Osp. Maggiore della Carità, Novara
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale di Piacenza, ASL Piacenza, Piacenza

REFERENCES:
- [Derived] Petracci E, Passardi A, Biggeri A, Valgiusti M, Monti M, Frassineti GL, Nanni O, Scarpi E. Baseline and Longitudinal Neutrophil-to-Lymphocyte Ratio as Prognostic Factor for Metastatic Colorectal Cancer: A Secondary Analysis of the ITACa Randomized Trial. JCO Precis Oncol. 2024 Jan;8:e2300256. doi: 10.1200/PO.23.00256. PMID 38295317
- [Derived] Casadei Gardini A, Scarpi E, Valgiusti M, Monti M, Ruscelli S, Matteucci L, Bartolini G, Vertogen B, Pagan F, Rovesti G, Frassineti GL, Passardi A. Prognostic role of a new index (multi inflammatory index) in patients with metastatic colorectal cancer: results from the randomized ITACa trial. Ther Adv Med Oncol. 2020 Sep 28;12:1758835920958363. doi: 10.1177/1758835920958363. eCollection 2020. PMID 33062063
- [Derived] Casadei-Gardini A, Scarpi E, Ulivi P, Palladino MA, Accettura C, Bernardini I, Spallanzani A, Gelsomino F, Corbelli J, Marisi G, Ruscelli S, Valgiusti M, Frassineti GL, Passardi A. Prognostic role of a new inflammatory index with neutrophil-to-lymphocyte ratio and lactate dehydrogenase (CII: Colon Inflammatory Index) in patients with metastatic colorectal cancer: results from the randomized Italian Trial in Advanced Colorectal Cancer (ITACa) study. Cancer Manag Res. 2019 May 10;11:4357-4369. doi: 10.2147/CMAR.S198651. eCollection 2019. PMID 31191000
- [Derived] Passardi A, Scarpi E, Tamberi S, Cavanna L, Tassinari D, Fontana A, Pini S, Bernardini I, Accettura C, Ulivi P, Frassineti GL, Amadori D. Impact of Pre-Treatment Lactate Dehydrogenase Levels on Prognosis and Bevacizumab Efficacy in Patients with Metastatic Colorectal Cancer. PLoS One. 2015 Aug 5;10(8):e0134732. doi: 10.1371/journal.pone.0134732. eCollection 2015. PMID 26244985
- [Derived] Passardi A, Nanni O, Tassinari D, Turci D, Cavanna L, Fontana A, Ruscelli S, Mucciarini C, Lorusso V, Ragazzini A, Frassineti GL, Amadori D. Effectiveness of bevacizumab added to standard chemotherapy in metastatic colorectal cancer: final results for first-line treatment from the ITACa randomized clinical trial. Ann Oncol. 2015 Jun;26(6):1201-1207. doi: 10.1093/annonc/mdv130. Epub 2015 Mar 3. PMID 25735317
- Available data/document: study publication — https://www.ncbi.nlm.nih.gov/pubmed/25735317 — Passardi A et al. Effectiveness of bevacizumab added to gold standard chemotherapy in metastatic colorectal cancer: final results of first-line from the ITACa randomized clinical trial. Ann Oncol 2015 Jun;26(6):1201-7
- Available data/document: study publication — https://www.ncbi.nlm.nih.gov/pubmed/26244985 — Passardi A et al. Impact of Pre-Treatment Lactate Dehydrogenase Levels on Prognosis and Bevacizumab Efficacy in Patients with Metastatic Colorectal Cancer. PLoS One 2015; 10(8): e0134732
- Available data/document: study publication — https://www.ncbi.nlm.nih.gov/pubmed/27120807 — Passardi A et al. Inflammatory indexes as predictors of prognosis and bevacizumab efficacy in patients with metastatic colorectal cancer. Oncotarget 2016 May 31;7(22):33210-9
- Available data/document: study publication — https://www.ncbi.nlm.nih.gov/pubmed/26259598 — Ulivi P et al. eNOS polymorphisms as predictors of efficacy of bevacizumab-based chemotherapy in metastatic colorectal cancer: data from a randomized clinical trial. J Transl Med 2015;11(3): 258
- Available data/document: study publication — https://www.ncbi.nlm.nih.gov/pubmed/26848624 — Casadei Gardini A et al. Prognostic role of serum concentrations of high-sensitivity C-reactive protein in patients with metastatic colorectal cancer: results from the ITACa trial. Oncotarget 2016 Mar 1;7(9):10193-202
- Available data/document: study publication — https://www.ncbi.nlm.nih.gov/pubmed/28465540 — Marisi G et al Circulating VEGF and eNOS variations as predictors of outcome in metastatic colorectal cancer patients receiving bevacizumab. Sci Rep 2017 May 2;7(1):1293